Date: 2025-08-31

**Unique Protocol ID: 2024-07566-01** 

Title: The Time Before the Crime - Risk Patterns in Offenders Undergoing a Forensic

**Psychiatric Evaluation (Tibec)** 

Principal Investigator: Katarina Howner, Associate professor, Karolinska Institutet

## Review Template: Variables for Review of Section 7 Examinations and Forensic Psychiatric Evaluations

| Variable | Outcome |
|---|---|
| Case number (Swedish National Board of Forensic Medicine) | |
| Date of review | |
| Reviewer (name) | |
| Criminal charge(s) (free text) | |
| Index offense, criminal charge (free text) | |
| Violent crime (including arson and robbery) | Yes□ No□ |
| Lethal violence (including manslaughter and attempted murder) | Yes □ No □ |
| Sexual offense | Yes□ No□ |
| Age at index offence | |
| Gender | Male □ Female □ |
| Previous convictions | Yes □ No □ |
| Previous entries in criminal record (number) | |
| Relationship with victim/complainant | Unknown □ Acquaintance □ Close relationship □ Family □ Partner □ |
| Modus operandi, in violent crime | Blunt force □ Knife □ Firearm □ Strangulation □ Other □ |
| Intoxication at the time of the offense | Drugs □ Alcohol □ Sober □ Unknown □ |

| Suicide attempt in connection with the offense | Yes □ No □ Unknown □ |
|---|---|
| Contact with psychiatric services | Ever □ Past month □ Past week □ Past 24 hours □ No □ Unknown □ |
| Primary diagnosis (free text) | |
| Secondary diagnosis/diagnoses (free text) | |
| Assessed to have a severe mental disorder (SMD) at the time of the offense | Yes □ No □ |
| Assessed to have SMD at the time of the evaluation | Yes □ No □ |
| Lacked capacity for insight and/or behavioral control | Yes □ Impaired □ No □ |
| Solid Violatico III de la contract | Not answered □ |
| Mental disorder not classified as severe | Yes □ No □ |
| District Court Ruling (free text) | |
| Court of Appeal Ruling (free text) | |

Note: SMD = Severe Mental Disorder (Swedish: Allvarlig Psykisk Störning)